CLINICAL TRIAL: NCT01208467
Title: Validating The Prognostic Role of ATR Mutation in Patients With Endometrioid Endometrial Cancer
Brief Title: Prognostic Biomarkers in Patients With Endometrial Cancer
Status: Completed | Type: Observational
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Other Study IDs: GOG-8017; NCI-2011-02870 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); GOG-8017; CDR0000685834; GOG-8017 (Other: Gynecologic Oncology Group); GOG-8017 (Other: CTEP); U10CA027469 (NIH)
Record Dates: First submitted 2010-09-23; First posted 2010-09-24 (Estimated); Last update posted 2017-08-23 (Actual); Status verified 2017-08

CONDITIONS: Endometrial Adenocarcinoma; Recurrent Uterine Corpus Carcinoma; Stage I Uterine Corpus Cancer; Stage II Uterine Corpus Cancer; Stage III Uterine Corpus Cancer; Stage IV Uterine Corpus Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Basic science (DNA analysis): DNA extracted from previously collected tumor samples is analyzed to validate the clinicopathologic associations and prognostic significance of ATR mutation.
  Interventions: Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This research study is studying prognostic biomarkers in tissue samples from patients with endometrial cancer. Studying samples of tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To validate the clinicopathologic associations and prognostic significance of ATR mutation in endometrioid endometrial cancer cases with defective DNA mismatch repair.

OUTLINE: This is a multicenter study.

DNA extracted from previously collected tumor samples is analyzed to validate the clinicopathologic associations and prognostic significance of ATR mutation.

ELIGIBILITY:
Inclusion Criteria:

* Women who were eligible and evaluable for the GOG-0210 molecular staging protocol in women with endometrial cancer

  * Women who were registered during the unrestricted enrollment period (through 9/23/07) will automatically qualify
  * Women who were registered during the restricted enrollment period (after 9/23/07) will only be considered if needed
* Women who had histologically confirmed endometrioid endometrial adenocarcinoma regardless of stage or grade
* Women who have defective DNA mismatch repair and are microsatellite instability positive (MSI+ and MSI-low)
* Women who consented to allow their specimens and clinical data to be used for future cancer research
* Women who have sufficient high-quality genomic DNA from tumor available for mutation analysis of ATR

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with endometrial cancer
Sampling Method: Non-Probability Sample
Enrollment: 2824 (Estimated)
Dates: Start 2010-09 (Actual); Primary Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
ATR mutation status | 1 month
  Parametric and non-parametric statistical tests will be performed to evaluate the association between ATR mutation status and demographic and clinical data. Product-limit estimates according to Kaplan-Meier method will be calculated and difference between survival according to ATR mutation status will be assessed using a two sided log rank test. The predictive ability of the final model will be assessed using a concordance index (C-statistic).
Microsatellite instability (MSI) | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Israel Zighelboim, Principal Investigator — Gynecologic Oncology Group
Locations (1):
- Gynecologic Oncology Group, Philadelphia, Pennsylvania, United States